CLINICAL TRIAL: NCT00492206
Title: A Phase II Study of Cetuximab in Combination With External Beam Radiation Followed By Consolidation Chemotherapy for Patients With Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Cetuximab With Radiation Followed by Consolidation Chemotherapy for NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Ahmad Tarhini, Associate Professor of Medicine and Translational Science, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-106; NCT00492206 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Non Small Cell Lung Cancer; NSCLC; EGFR Inhibitor; Radiation Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): Cetuximab 400 mg/m2 IV week 0 only
  External beam radiation weeks 1 - 7
  Cetuximab 250 mg/m2 IV weekly thereafter weeks 1 - 7
  Cetuximab 250 mg/m2 IV weekly weeks 8 - 26
  Carboplatin AUC = 6 IV Paclitaxel 200 mg/m2 IV Every 3 weeks x 3 Cycles
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — The initial dose of cetuximab is 400 mg/m2 intravenously administered over 120 minutes, followed by weekly infusions at 250 mg/m2 IV over 60 minutes. Subjects will receive cetuximab from week 0 through week 26.
  Other Names: Erbitux, C225

SUMMARY:
This is an open label, phase II study in which cetuximab with concurrent thoracic radiotherapy followed by consolidation chemotherapy with paclitaxel/carboplatin/cetuximab will be administered to subjects with locally advanced NSCLC.

DETAILED DESCRIPTION:
This is a Phase II study to determine the overall survival for patients with locally advanced NSCLC treated with cetuximab with concurrent thoracic radiotherapy followed by consolidation chemotherapy with paclitaxel/carboplatin/cetuximab. This is a multicenter study including 36 subjects who will be males and females, both greater than 18 years of age. All subjects will initially receive radiation and cetuximab. Radiation will be given once a day (Monday-Friday) for approximately 6-8 weeks. During the course of radiation, cetuximab will be given intravenously once a week. Approximately 4-6 weeks after the last radiation dose, the subjects will be treated with chemotherapy, paclitaxel/carboplatin. Chemotherapy will be given intravenously once every 3 weeks for 3 cycles (1 cycle=3 weeks). Cetuximab intravenous administration will be continued throughout the entire study, once a week through week 26 including during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of non-small cell lung cancer
* Patients must have surgically unresectable stage IIIA disease or stage IIIB disease without malignant pleural/pericardial effusion
* Patients must have measurable disease as per the RECIST criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 9.2 for the evaluation of measurable disease.
* Age >18 years. Lung cancer is extremely rare in children.
* ECOG performance status 0-1 (Karnofsky >70%; see Appendix A).
* If available, tumor tissue should be submitted for EGFR status by IHC and correlative studies.
* Patients must have normal organ and marrow function as defined below:
* leukocytes >3,000/μL
* absolute neutrophil count >1,500/μL
* platelets >100,000/μL
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* The effects of cetuximab on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because EGFR inhibitors, chemotherapeutic agents and radiation therapy, as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Willingness to sign an approved informed consent.

Exclusion Criteria:

* Patients should not have received prior chest radiation therapy.
* Patients with a history of pulmonary fibrosis are excluded from study.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, paclitaxel, cetuximab or other agents used in the study.
* History of any cancer other than NSCLC (except non-melanoma skin cancer or carcinoma in situ of the cervix) within the last five years.
* Prior therapy with known specific inhibitors of the EGFR.
* History of severe allergic reaction to prior therapy with monoclonal antibodies
* Peripheral neuropathy of more than grade 1 in severity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, significant history of uncontrolled cardiac disease ie. uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure,and cardiomyopathy with decreased ejection fraction, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because carboplatin, paclitaxel, cetuximab and radiation therapy have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the above agents, breastfeeding should be discontinued if the mother is treated with the agents used in this study. These potential risks may also apply to other agents used in this study.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with carboplatin, paclitaxel and cetuximab or other agents administered during the study. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Active hepatitis.
* History of pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Principal Investigator — University of Pittsburgh
Locations (31):
- United States (31):
  - Sylvester Comprehensive Cancer Center, University of Miami, Miami, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - UPMC Cancer Center -Teramana Cancer Center, Steubenville, Ohio
  - UPMC Cancer Center -Beaver, Beaver, Pennsylvania
  - UPMC Cancer Center - Clairton, Clairton, Pennsylvania
  - UPMC Cancer Center - Oakbrook Commons, Greensburg, Pennsylvania
  - UPMC Cancer Center -Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Cancer Institute, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Center -Indiana, Indiana, Pennsylvania
  - UPMC Cancer Center -John P. Murtha Pavilion, Johnstown, Pennsylvania
  - UPMC Cancer Center -McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center -Haymaker Rd., Monroeville, Pennsylvania
  - UPMC Cancer Center -Mosside Blvd., Monroeville, Pennsylvania
  - UPMC Cancer Center -Sewickley Medical Center, Moon Township, Pennsylvania
  - UPMC Cancer Center -Mt. Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Cancer Center -Jameson, New Castle, Pennsylvania
  - UPMC Cancer Center -New Castle, New Castle, Pennsylvania
  - UPMC Presbyterian -Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -Delafield Rd., Pittsburgh, Pennsylvania
  - UPMC Cancer Center -St. Margaret, Pittsburgh, Pennsylvania
  - Universtity of Pittsburgh Cancer Institute -Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -Drake, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -St. Clair, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center -Robert Eberly Pavilion, Uniontown, Pennsylvania
  - UPMC Cancer Center -Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center -Washington, Washington, Pennsylvania
  - UPMC Cancer Center -Wexford, Wexford, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from the surgically unresectable stage IIIA or IIIB NSCLC patient populations
Pre-assignment Details: Non-Small Cell Lung Cancer, unresectable limited to Stage IIIA/B.
Groups:
- Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca: Participants (with surgically unresectable stage IIIA or IIIB NSCLC) received Cetuximab 400 mg/m2 IV (week 0 only), External beam radiation (weeks 1 - 7) and Cetuximab 250 mg/m2 IV weekly thereafter (weeks 1 - 7). Weeks 4-6 was the pre-consolidation phase during which participants received Carboplatin AUC = 6 IV, Paclitaxel 200 mg/m^2 IV Every 3 weeks x 3 Cycles. Cetuximab was given for up to a total of 26 weeks.
Period: Overall Study
Arm/Group | Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of patients with surgically unresectable stage IIIA or IIIB NSCLC accrued
Arm/Group | Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] — Age greater than or equal to 18 years of age
  years | 67 [40 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Time Frame: Up to 36 months
Population: Patients with surgically unresectable stage IIIA or IIIB NSCLC. Survival analysis excluded the two ineligible patients with advanced NSCLC (N = 38).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Received ≥1 Dose of Cetuximab: Participants (with surgically unresectable stage IIIA or IIIB NSCLC) received Cetuximab 400 mg/m2 IV (week 0 only), External beam radiation (weeks 1 - 7) and Cetuximab 250 mg/m2 IV weekly thereafter (weeks 1 - 7). Weeks 4-6 was the pre-consolidation phase during which participants received Carboplatin AUC = 6 IV, Paclitaxel 200 mg/m^2 IV Every 3 weeks x 3 Cycles. Cetuximab was given for up to a total of 26 weeks.
Arm/Group | Received ≥1 Dose of Cetuximab
Number analyzed (Participants) | 38
months | 19.4 [15.4 to 26]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Response and progression were evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]. Progressive Disease was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 36 months
Population: Patients with surgically unresectable stage IIIA or IIIB NSCLC. Survival analysis excluded the two ineligible patients with advanced NSCLC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Received ≥1 Dose of Cetuximab
Number analyzed (Participants) | 38
months | 9.3 [8.5 to 17.2]

3. Secondary Outcome: Best Overall Response Rate (ORR) (Number of Participants)
Description: The Best Overall Response is the best response (Complete Response, Partial Response, Stable Disease, Progressive Disease) recorded from the start of the study treatment until the disease progression/recurrence at end of study. Response and progression were evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]. Complete Response (CR) is the Disappearance of all target lesions and Partial Response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks after treatment initiation
Population: Patients who received concurrent radiotherapy + cetuximab + consolidation therapy, and patients who did not receive cetuximab
Measure: Number; unit: participants
Groups:
- Received Concurrent Radiotherapy + Cetuximab: Participants (with surgically unresectable stage IIIA or IIIB NSCLC) received Cetuximab 400 mg/m2 IV (week 0 only), External beam radiation (weeks 1 - 7) and Cetuximab 250 mg/m2 IV weekly thereafter (weeks 1 - 7). Weeks 4-6 was the pre-consolidation phase during which participants received Carboplatin AUC = 6 IV, Paclitaxel 200 mg/m^2 IV Every 3 weeks x 3 Cycles. Cetuximab was given for up to a total of 26 weeks.
Arm/Group | Received Concurrent Radiotherapy + Cetuximab
Number analyzed (Participants) | 40
participants
  Complete Response (CR) Rate | 4
  Partial Response (PR) Rate | 18
  Stable Disease | 4
  Progressive Disease | 6
  Not evaluable | 8

4. Secondary Outcome: EGFR (Epidermal Growth Factor Receptor) Gene Mutation and Akt, pAkt, and MAPKinase
Description: EGFR (epidermal growth factor receptor) gene mutation status and Akt, pAkt, and MAPKinase in participant tumor tissue.
Time Frame: approx. 5 years
Population: Participants with baseline tumor tissue available for EGFR status analysis by fluorescence in situ hybridization (FISH). Akt, pAkt, and MAPKinase analyses were not conducted.
Measure: Number; unit: percentage of tumors
Units Other Than Participants: baseline tumor tissue
Arm/Group | Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca
Number analyzed (Participants) | 26
Number analyzed (baseline tumor tissue) | 26
percentage of tumors | 65

ADVERSE EVENTS:
Description: Adverse events (AEs) include all AEs (those considered related or unrelated to study treatment)
Arm/Group | Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca
Serious Adverse Events (participants affected / at risk) | 11/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca (N=40)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Hypotension (Cardiac disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Muscle weakness, generalized or specific area (not due to neuropathy), Extraocular (Musculoskeletal and connective tissue disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8
Pain, Abdomen NOS (General disorders) | 2
Rigors/chills (General disorders) | 1
Supraventricular and nodal arrhythmia, Atrial fibrillation (Cardiac disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chest Radiotherapy + Cetuximab + Consolidation Therapy With ca (N=40)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 20
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 24
Supraventricular and nodal arrhythmia, Atrial fibrillation (Cardiac disorders) | 3
Supraventricular and nodal arrhythmia, Sinus tachycardia (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 4
Constitutional Symptoms - Other (Specify, __) (General disorders) | 4
Sweating (diaphoresis) (General disorders) | 4
Rigors/chills (General disorders) | 6
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 8
Insomnia (General disorders) | 8
Weight loss (General disorders) | 11
Fatigue (asthenia, lethargy, malaise) (General disorders) | 29
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Nail changes (Skin and subcutaneous tissue disorders) | 4
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 8
Rash: dermatitis associated with radiation, Radiation (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 11
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 31
Hemorrhoids (Gastrointestinal disorders) | 3
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 6
Heartburn/dyspepsia (Gastrointestinal disorders) | 6
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 10
Esophagitis (Gastrointestinal disorders) | 11
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 14
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 16
Anorexia (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 23
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 3
Infection - Other (Specify, __) (Infections and infestations) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 5
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 6
Mood alteration, Depression (Nervous system disorders) | 3
Neurology - Other (Specify, __) (Nervous system disorders) | 3
Neuropathy: motor (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 4
Mood alteration, Anxiety (Nervous system disorders) | 4
Syncope (fainting) (Nervous system disorders) | 6
Neuropathy: sensory (Nervous system disorders) | 13
Dry eye syndrome (Eye disorders) | 3
Watery eye (epiphora, tearing) (Eye disorders) | 3
Pain - Other (Specify, __) (General disorders) | 3
Pain, Abdomen NOS (General disorders) | 3
Pain, Throat/pharynx/larynx (General disorders) | 3
Pain, Chest/thorax NOS (General disorders) | 4
Pain, Muscle (General disorders) | 4
Pain, Bone (General disorders) | 5
Pain, Extremity-limb (General disorders) | 5
Pain, Joint (General disorders) | 5
Pain, Back (General disorders) | 6
Pain, Head/headache (General disorders) | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 6
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 31
Thrombosis/thrombus/embolism (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less